CLINICAL TRIAL: NCT05605847
Title: Adherence of Imaging Order to the 2020 French Guidelines for Patients With Cervical Spine Injury in the Emergency Setting: a Retrospective Cohort Study
Brief Title: Adherence of Imaging Order to the 2020 French Guidelines for Patients With Cervical Spine Injury in the Emergency Setting
Acronym: MINERVA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MINERVA
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Cervical Spine Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cervical spine trauma is a frequent reason for consultation in emergency medicine. It concerns approximately 10,000 patients admitted to the emergency room each year in France. There are two types of cervical spine trauma: penetrating and non-penetrating. Non-penetrating injuries are the most frequent and can be classified according to the mechanism involved. Whiplash is the most common type of trauma in emergency medicine. The injuries associated with this type of trauma predominate in the mobile spinal segment and are most often benign: only 2 to 3% of conscious patients consulting the emergency room actually present with cervical injuries such as fractures, dislocations or unstable sprains. In emergency medicine, the paradigm is therefore to identify patients at risk of complications, minimizing the need for unnecessary and radiating imaging. Although cervical spine trauma is a frequent reason for emergency room visits, the incidence of anatomical lesions is generally low and the X-rays prescribed most often do not show any abnormality. For cervical lesion screening to be safe and effective, the screening rules must have a high sensitivity, a low negative likelihood ratio, and a low false positive rate. Two clinical prediction rules have been extensively evaluated in the literature to guide imaging for nonpenetrating cervical injuries: the National Emergency X-Radiography Utilization Study (NEXUS) rule and the Canadian C-Spine 5 rule. The NEXUS rule4 applies to any clinically stable patient (Glasgow Coma Scale 15, systolic blood pressure ≥ 90 mmHg, and respiratory rate between 10 and 24/min) presenting to the emergency department with a nonpenetrating trauma. The criteria constituting the NEXUS clinical rule are:

* Absence of tenderness on palpation of the posterior cervical midline ;
* Normal state of alertness (Glasgow Coma Scale 15);
* Absence of focal neurological deficit;
* Absence of signs of intoxication;
* Absence of distracting pain (other pain that may mask neck pain, e.g., long bone fracture).

If these 5 criteria are present, the risk of cervical spine injury is low and no imaging is recommended.

The Canadian C-Spine 5 rule applies to patients who are 16 years of age or older; conscious with a Glasgow Coma Scale of 15; stable (systolic blood pressure ≥ 90 mmHg and respiratory rate between 10 and 24/min); and have had head or neck trauma in the past 48 hours. As soon as the rules of clinical prediction do not make it possible to rule out the hypothesis of a spinal injury, the exploration of cervical trauma traditionally involves the performance of radiographic images. They must include the following incidences: face, profile and open mouth centered on the cervico-occipital hinge ("open mouth odontoid"). Nevertheless, the sensitivity of these conventional radiographs for the detection of cervical spine lesions is poor, about 50%. Thus, the use of standard radiographs is usually limited to conscious, ambulatory patients at low risk of spinal injury. Conversely, the cervical CT is the reference examination for the detection of spinal bone lesions with a sensitivity close to 100%. Its sensitivity is superior to that of radiographic images in both high-risk and low-risk patients with spinal injuries. Difficulty of access and exposure to ionizing radiation, which is lower with standard radiography, generally influence the choice of imaging in the emergency room. In December 2020, the French High Authority for Health published a sheet on the relevance of cervical imaging in the context of non-penetrating cervical trauma. This sheet proposes a practical table according to the precise clinical context of the patient as well as the best first-line imaging. These good practice recommendations were part of an approach to improve the relevance of care. Cervical spine imaging for patients admitted to the emergency department for non-penetrating cervical spine trauma was recommended in one of the following situations

* patient 65 years of age or older ;
* patient unstable or with consciousness disorders or neurological signs;
* imaging recommended by one of the following two rules: NEXUS or Canadian C-Spine;
* a history of ankylosing spine (ankylosing spondylitis, hyperostosis, etc.), even in case of "minor" trauma;
* if a cervical artery dissection is suspected. Investigator's hypothesis is that the HAS recommendations of good cervical imaging practices for non-penetrating cervical trauma are difficult to apply routinely in emergency departments for several reasons: the frequency of consultations for cervical trauma, the limited availability of emergency CT scans, and the fear of radiation and unnecessary additional costs in emergency situations. Investigators wish to determine the actual rate of application of the clinical rules recommended by the HAS in the GHPSJ emergency department and the factors predicting their non-application by the GHPSJ team of emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient consulting the GHPSJ emergency department for a non-penetrating cervical spine injury from 01/01/2021 to 12/31/2021
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient consulting the GHPSJ emergency department for a non-penetrating cervical spine injury from 01/01/2021 to 12/31/2021
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with non-penetrating cervical trauma in the emergency department for whom there is a lack of compliance with the cervical spine imaging order | Day1
  This outcome corresponds to the proportion of patients for whom cervical spine imaging does not correspond to that recommended by the HAS strategy.

SECONDARY OUTCOMES:
Level of knowledge of emergency physicians on HAS recommendations | Day1
  This outcome corresponds to the percentage of physicians who provided at least 80% of responses to the questionnaire in agreement with the 2020 HAS recommendations.
Questionnaire of difficulties faced by emergency physicians in the management of whiplash injuries | Day1
  This outcome corresponds to the difficulties reported by emergency physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Camille NUSSBAUM, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Cusick JF, Yoganandan N. Biomechanics of the cervical spine 4: major injuries. Clin Biomech (Bristol). 2002 Jan;17(1):1-20. doi: 10.1016/s0268-0033(01)00101-2. PMID 11779642
- [Background] Pimentel L, Diegelmann L. Evaluation and management of acute cervical spine trauma. Emerg Med Clin North Am. 2010 Nov;28(4):719-38. doi: 10.1016/j.emc.2010.07.003. PMID 20971389
- [Background] Griffith B, Bolton C, Goyal N, Brown ML, Jain R. Screening cervical spine CT in a level I trauma center: overutilization? AJR Am J Roentgenol. 2011 Aug;197(2):463-7. doi: 10.2214/AJR.10.5731. PMID 21785095
- [Background] Hoffman JR, Mower WR, Wolfson AB, Todd KH, Zucker MI. Validity of a set of clinical criteria to rule out injury to the cervical spine in patients with blunt trauma. National Emergency X-Radiography Utilization Study Group. N Engl J Med. 2000 Jul 13;343(2):94-9. doi: 10.1056/NEJM200007133430203. PMID 10891516